CLINICAL TRIAL: NCT00924690
Title: Disparities in Colorectal Cancer Prevention Behaviors
Brief Title: Colon Cancer Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Lucia Leone, UNC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UNC-CCEP
Record Dates: First submitted 2009-04-06; First posted 2009-06-19 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Colorectal Cancer
Keywords: Colon; Cancer; Screening; Prevention; Information
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Behavioral Message Arm
  Interventions: Other: Behavioral Messages
- 2 (Active Comparator): Generic Message Arm
  Interventions: Other: Generic Messages

INTERVENTIONS:
Other: Behavioral Messages — Participants will read 10 behavioral messages about colon cancer screening and physical activity.
  Arms: 1
Other: Generic Messages — Individuals will read 10 generic messages about colon cancer screening and physical activity.
  Other Names: Control
  Arms: 2

SUMMARY:
The goal of this research study is to design messages which can help people learn more about how to prevent colon cancer. Eligible participants will be asked to review a series of short cancer prevention messages and share their opinions on them. Participants also need to fill out a short survey with questions on their background and attitudes and knowledge about physical activity and colon cancer. The whole study can be completed online and will take less than 1 hour. After completing the entire study, participants will receive $25.

If you are interested in participating in this study, please visit the following website:

https://surveys.chaicore.com/preventcancer/

DETAILED DESCRIPTION:
The goal of this research is to develop and test potential intervention messages which can be used to help increase colon cancer prevention behaviors. Two sets of intervention messages will be developed: generic and behavioral. Using a randomized control design the investigators will evaluate the behavioral messages among women. This message testing protocol will help them determine if the messages are relevant, acceptable, comprehensible, memorable, and motivating for the target audience. The investigators' hypothesis is that the behavioral messages will receive more positive ratings than the generic messages. If so, they will be used to promote cancer screening and physical activity in future intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 50-80 years old

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Elaboration using the Elaboration Likelihood Scale | This study is to be completed in one session. The outcome is measured immediately after reading messages

SECONDARY OUTCOMES:
Behavioral Intention to Engage in Colorectal Cancer Screening or Physical Activity | This study is to be completed in one session. The outcome is measured immediately after reading messages

CONTACTS AND LOCATIONS:
Overall Officials: Lucia A Leone, BA, Principal Investigator — UNC; Marci K Campbell, PhD, Study Chair — UNC
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States